CLINICAL TRIAL: NCT05454176
Title: Diabetes in African Youth: Improving Glucose Time-In-Range (DAYTime, Randomized Clinical Trial)
Brief Title: Diabetes in African Youth
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEDS-2022-31031
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: type1diabetes
Keywords: Uganda; type 1 diabetes; continuous glucose monitor; CGM; resource poor nations
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: randomized, non-blinded, phase 4 clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Libre 2 (Experimental): Half of patients will be randomized to wear an unblinded FreeStyle Libre 2 CGM for 12 months. Sensor glucose data will be continuously available to patients and their providers.
  Primary outcome measurement occurs at 6 months.
  Interventions: Device: Libre 2
- SMBG levels 3x/daily (standard diabetes management) (Placebo Comparator): Half of subjects will be given sufficient test strips to test 3x per day for the first 6 months of the study, as is usual clinical practice. They wear a blinded FreeStyle Libre Pro CGM monthly during this time-the blinded device is simply to collect study data, the data will not be available to the patient or their provider for clinical use. They will use the 3x daily SMBG data for insulin adjustment, as per usual standard of care. For the final 6 months (7-12), this group will switch to unblinded CGM patients and providers will have full access to CGM data.
  Interventions: Device: Device for SMBG and Libre Pro

INTERVENTIONS:
Device: Libre 2 — The unblinded FreeStyle Libre 2 CGM will be placed every two weeks during months 0-12 for the CGM Cohort. Patients will be taught to insert the sensor themselves.
  They will be given a 1 month supply at each monthly clinic visit and extra sensors in case a sensor falls out early. Patients will be given SMBG test strips to test capillary glucose for confirmation of any CGM glucose level <=60mg/dl. They will keep track of the number of times this is necessary. Patients will return used sensors at each clinic visit. The study team will upload the data to a study website. Patients and care providers will have access to unblinded sensor data for clinical use.
  Arms: Libre 2
Device: Device for SMBG and Libre Pro — A glucose meter and sufficient teststrips for fingerpoke glucose monitoring 3x/day will be provided for months 1-6. This is standard-of-care in Uganda. Glucose meters will be downloaded monthly in clinic as per usual clinical practice.
  DeviceBlinded CGM device: Libre Pro (blinded data collection device, not an intervention) The blinded FreeStyle Libre Pro CGM will be inserted at each monthly clinic visit to provide control data, months 0-6 for the Control Group. They will return all used sensors at each clinic visit. The study team will upload the data to a study website. Neither patients nor the local research teams will have access to the blinded sensor data for clinical use until the end of months 0-6 so as not to influence standard diabetes management. They will instead rely on SMBG values as per usual routine.
  After the first 6 months they will receive Libre 2 CGM systems as described above for the intervention group.
  Arms: SMBG levels 3x/daily (standard diabetes management)

SUMMARY:
This RCT aims to improve T1D care in East African children and young adults by testing the hypothesis that enabling patients to continuously monitor glucose levels with flash CGM technology will improve glucose time-in-range (glucose level 70-180 mg/dl). A second primary endpoint is to perform a cost analysis on flash glucose monitoring compared to 3x/day SMBG, to determine whether this technology is cost-effective in the setting of a less-resourced nation.

After a 2 week assessment with blinded CGM when a potential subject's ability to wear CGM is confirmed, subjects will be enrolled for 12 months in randomized, open label study, with a primary endpoint measurement at 6 months. All subjects will receive monthly diabetes self-management education.

For the first six months, months 1-6:

* Half of patients (n=90) will be randomized to an unblinded FreeStyle Libre 2 CGM.They and their care providers will be able to continuously see their CGM glucose levels to assist in insulin adjustment.
* Half of patients (n=90) will be given sufficient test strips for 3x daily SMBG while wearing blinded CGM (control group). Neither they nor their care providers will be able to see their CGM glucose levels (the blinded CGM is simply for outcome measurement, not an intervention). As per usual clinical practice, only the SMBG glucose levels will be available to assist in insulin adjustment.
* The change between baseline to 6 months in CGM-derived glucose percent time-in- range will be compared between groups (first primary study endpoint).

For the second six months, months 7-12:

* The control group will switch to unblinded CGM months 7-12 (their data months 7-12 months will be compared to their data months 1-6 as part of the primary endpoint assessment).
* The patients who wore the unblinded CGM months 1-6 will continue for another 6 months to assess the impact of wearing the CGM for 12 continuous months (a secondary endpoint).

Once the clinical portion of the study is complete, study investigators who are health economists from the Uganda Ministry of Health will perform a costs analysis (second primary endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Children and youth in Uganda, age 4-26 years at the beginning of the baseline assessment
* T1D (determined by clinical criteria, as autoantibody testing is not regionally available) of at least 12 months duration at the beginning of the baseline assessment
* Receiving insulin therapy
* Access to a cell phone (nearly ubiquitous in Uganda, even in remote areas)
* At least one parent or guardian (or as per local regulations) is present in clinic and able to give consent for children under 18 years of age (those age 18-26 may give consent for themselves)

Exclusion Criteria:

* Unwilling or unable to be seen monthly at the pediatric diabetes clinic
* Pregnant or breast-feeding; women likely to become pregnant in the next year
* Major medical conditions which the investigator feels would interfere with study participation
* Patient already has CGM
* Inability during the baseline assessment period to wear the sensor for at least 7 days or return it
* Participant deemed unlikely or unable to comply with the protocol

Ages: 4 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2027-08-15 (Estimated); Study Completion 2027-08-15 (Estimated)

PRIMARY OUTCOMES:
Glucose Time-in-Range | 6 months
  The change in glucose Time-in-Range (percent time glucose levels are 70-180 mg/dl) from baseline to six months will be compared between patients wearing the unblinded CGM to those performing standard 3x/day SMBG.
Cost analysis of CGM | 1 year
  Cost analysis on flash glucose monitoring compared to 3x/day SMBG, to determine whether this technology is cost effective in the setting of a low-resource nation.

CONTACTS AND LOCATIONS:
Overall Officials: Antoinette Moran, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States